CLINICAL TRIAL: NCT00206128
Title: 6-week Multicenter, Double-blind, Randomized, Parallel-group, Phase 3 Study to Evaluate the Feasibility of Switching From Immediate-release Quetiapine Fumarate (SEROQUEL) to Sustained-release Quetiapine Fumarate in Outpatients With Schizophrenia (Abbreviated)
Brief Title: Immediate Release (IR) to Sustained Release (SR) Switching Study: Study of Switching From IR Seroquel to SR Seroquel in Outpatients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1444C00146
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Seroquel SR

SUMMARY:
The purpose of this study is to determine that the efficacy of the sustained release (SR) formulation of quetiapine (Seroquel) is not inferior to the immediate release (IR) formulation.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* A stable dose of quetiapine IR between 300 and 800 mg/day within 4 weeks prior to the enrolment visit (Visit 1) as judged by the investigator.
* Female patients of childbearing potential must have a negative serum pregnancy test at enrolment and be willing to use a reliable method of birth control, ie, barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal ligation during the study.
* Able to understand and comply with the requirements of the study, as judged by the investigator.

Exclusion Criteria:

* Meeting the criteria for any other (than schizophrenia) Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) Axis I diagnosis, concomitant organic mental disorder or mental retardation.
* Patients with substance abuse or dependence, as defined by DSM-IV, and not in full remission. A urine drug screen test will be performed. The investigator will evaluate the results along with medical history to determine if the patient meets DSM-IV criteria for substance abuse or dependence.
* Risk of transmitting human immunodeficiency virus (HIV) or hepatitis B, via blood or other body fluids, as judged by the investigator.
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2004-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who discontinue study treatment due to lack of efficacy or whose positive and negative syndrome scale (PANSS) total score increases 20% or more | from randomisation to any visit

SECONDARY OUTCOMES:
The change in PANSS total score | from randomization to week 6
The change in PANSS positive, negative and general psychopathology symptoms subscale scores respectively | from randomization to week 6
The proportion of patients with a Clinical Global Impressions - Improvement (CGI-I) score greater than or equal to 4 | at week 6

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (69):
- United States (18):
  - Research Site, Birmingham, Alabama
  - Research Site, Anaheim, California
  - Research Site, Cerritos, California
  - Research Site, Garden Grove, California
  - Research Site, National City, California
  - Research Site, Pasadena, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, North Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Hoffman Estates, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Jackson, Mississippi
  - Research Site, Clementon, New Jersey
  - Research Site, Staten Island, New York
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
- Research Site, QLD, Australia
- Bulgaria (3):
  - Research Site, Burgas
  - Research Site, Radnevo
  - Research Site, Varna
- Canada (9):
  - Research Site, Vancouver, British Columbia
  - Research Site, Aurora, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Orléans, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Prince Albert, Saskatchewan
- Estonia (3):
  - Research Site, Põltsamaa
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Mikkeli
  - Research Site, Turku
- Germany (7):
  - Research Site, München, Bavaria
  - Research Site, Göttingen, Lower Saxony
  - Research Center, Aachen, North Rhine-Westphalia
  - Research Site, Aachen, North Rhine-Westphalia
  - Research Site, Jena, Thuringia
  - Research Site, Halle
  - Research Site, Marburg
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Nagykálló
  - Research Site, Szeged
  - Research Site, Székesfehérvár
- Italy (7):
  - Research Site, Bologna, BO
  - Research Site, Cagliari, CA
  - Research Site, Città di Castello, PG
  - Research Site, Ellera Di Corciano, PG
  - Research Site, Torino, TO
  - Research Site, Bassano del Grappa, VI
  - Research Site, Quartu Sant'Elena
- Latvia (2):
  - Research Site, Riga
  - Research Site, Sigulda
- Lithuania (4):
  - Research Site, Ziegzdrai, Kaunas County
  - Research Site, Klapeda
  - Research Site, Šiauliai
  - Research Sitte, Vilnius
- Spain (6):
  - Research Site, Jerez de la Frontera, Cádiz
  - Research Site, Alcobendas, Madrid
  - Research Site, Colmenar Viejo, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Móstoles, Madrid
  - Research Site, Villamartín